CLINICAL TRIAL: NCT02219490
Title: An Open-Label, Multicenter Study to Evaluate Long-Term Outcomes With ABT-450/Ritonavir/ ABT-267 (ABT-450/r/ABT-267) and ABT-333 With or Without Ribavirin (RBV) in Adults With Genotype 1 Chronic Hepatitis C Virus (HCV) Infection (TOPAZ-I)
Brief Title: A Study to Evaluate Long-term Outcomes Following Treatment With ABT-450/Ritonavir/ABT-267 (ABT-450/r/ABT-267) and ABT-333 With or Without Ribavirin (RBV) in Adults With Genotype 1 Chronic Hepatitis C Virus (HCV) Infection
Acronym: TOPAZ-I
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M14-423; 2014-001022-14 (EudraCT Number)
Record Dates: First submitted 2014-08-15; First posted 2014-08-19 (Estimated); Results first posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2022-06

CONDITIONS: Chronic Hepatitis C Virus (HCV) Infection Genotype 1
Keywords: Hepatitis C Genotype 1; Compensated Cirrhosis; Cirrhosis; Naive; Hepatitis C; Hepatitis C Virus; Treatment-Experienced; Relapser; Null responder; Non responder
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C; Fibrosis | interventions — paritaprevir; ombitasvir; dasabuvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ABT-450/r/ABT-267 plus ABT-333 with or without ribavirin (RBV) (Experimental): Participants with HCV GT1b without cirrhosis received the 3-DAA (ABT-450/ritonavir/ABT-267 and ABT-333) regimen: two 75 mg ABT-450/50 mg ritonavir/12.5 mg ABT-267 tablets taken orally every morning (QD) and one ABT-333 250 mg tablet taken orally twice a day (BID) for 12 weeks. Participants with HCV GT1a without cirrhosis and those with HCV GT1b with cirrhosis received the 3-DAA regimen and weight-based ribavirin (RBV; 1000 to 1200 mg divided twice daily per local label) for 12 weeks. Participants with HCV GT1a with cirrhosis received the 3-DAA regimen and weight-based RBV per local label for 24 weeks.
  Interventions: Drug: ABT-450/r/ABT-267; Drug: ABT-333; Drug: Ribavirin (RBV)

INTERVENTIONS:
Drug: ABT-450/r/ABT-267 — Tablet for oral use
  Other Names: ABT-450 also known as paritaprevir; ABT-267 also known as ombitasvir; Paritaprevir/ritonavir/ombitasvir also known as Viekirax
Drug: ABT-333 — Tablet for oral use
  Other Names: ABT-333 also known as dasabuvir; ABT-333 also known as Exviera
Drug: Ribavirin (RBV) — Ribavirin was provided as 200 mg tablets, and dosed based on weight,1000 to 1200 mg divided twice daily per local label. For example, for participants weighing < 75 kg, RBV may have been taken orally as 2 tablets in the morning and 3 tablets in the evening which corresponds to a 1000 mg total daily dose. For participants weighing ≥ 75 kg, RBV may have been taken orally as 3 tablets in the morning and 3 tablets in the evening which corresponds to a 1200 mg total daily dose.

SUMMARY:
The purpose of this study was to evaluate the effect of treatment with ABT-450 co-formulated with ritonavir and ABT-267 (ABT-450/r/ABT-267) and ABT-333; 3-DAA regimen, with or without ribavirin (RBV) in adults with chronic hepatitis C virus genotype 1 (HCV GT1) infection.

DETAILED DESCRIPTION:
This study (TOPAZ-I; M14-423), was a Phase 3b, open-label, multicenter study conducted outside of the United States which, together with its companion study TOPAZ-II (M14-222; NCT 02167945) conducted in the United States, was designed with the primary objective of assessing the effect of treatment response on long-term clinical outcomes in adults with chronic HCV GT1 infection with or without compensated cirrhosis, who were either treatment-naïve or interferon/ribavirin (IFN/RBV) treatment- experienced. In both studies, participants were treated with the 3-DAA regimen with or without RBV. This study consisted of a screening period of up to 42 days, a treatment period of either 12 weeks for HCV GT1a-infected subjects without cirrhosis and for HCV GT1b-infected subjects without cirrhosis or with compensated cirrhosis or 24 weeks for GT1a-infected participants with compensated cirrhosis, and a 260-week post-treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females at least 18 years old at screening
2. Females must be post-menopausal for more than 2 years or surgically sterile or practicing acceptable forms of birth control
3. Chronic hepatitis C, genotype 1 infection
4. Males must be surgically sterile or agree to practice acceptable forms of birth control
5. Screening laboratory result indicating HCV genotype 1 infection

Exclusion Criteria:

1. Use of contraindicated medications within 2 weeks of dosing
2. Abnormal laboratory tests
3. Current or past clinical evidence of Child-Pugh B or C classification or history of liver decompensation
4. Confirmed presence of hepatocellular carcinoma
5. History of solid organ transplant

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1596 (Actual)
Dates: Start 2014-10-30 (Actual); Primary Completion 2021-05-13 (Actual); Study Completion 2021-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (187):
- Algeria (3):
  - CHU Bab El Oued /ID# 145420, Algiers
  - CHU Bologhine Hospital /ID# 145421, Algiers
  - CHU Mustapha Bacha /ID# 132130, Algiers
- Australia (8):
  - St Vincent's Hospital Sydney /ID# 131001, Darlinghurst, New South Wales
  - Nepean Hospital /ID# 130999, Kingswood, New South Wales
  - Westmead Hospital /ID# 130997, Westmead, New South Wales
  - Greenslopes Private Hospital /ID# 131003, Greenslopes, Queensland
  - Royal Brisbane and Women's Hospital /ID# 131004, Herston, Queensland
  - Royal Adelaide Hospital /ID# 131002, Adelaide, South Australia
  - St Vincent's Hospital Melbourne /ID# 131000, Fitzroy Melbourne, Victoria
  - The Royal Melbourne Hospital /ID# 130998, Parkville, Victoria
- Austria (3):
  - Medizinische Universitaet Graz /ID# 131018, Graz, Styria
  - Ordensklinikum Linz GmbH Elisabethinen /ID# 131017, Linz, Upper Austria
  - Medizinische Universitaet Wien /ID# 131015, Vienna, Vienna
- Belgium (3):
  - Cliniques Universitaires de Bruxelles Hopital Erasme /ID# 131020, Brussels, Brussels Capital
  - UCL Saint-Luc /ID# 131019, Woluwe-Saint-Lambert, Brussels Capital
  - Universitair Ziekenhuis Leuven /ID# 131021, Leuven, Vlaams-Brabant
- Bulgaria (5):
  - Tokuda Hospital Sofia /ID# 131022, Sofia
  - UMHAT Sveti Ivan Rilski /ID# 131026, Sofia
  - Univ Hosp for Active Treat /ID# 131023, Sofia
  - Diagnostic Consultative Center /ID# 131027, Sofia
  - UMHAT Sveta Marina /ID# 131025, Varna
- Canada (15):
  - University of Calgary /ID# 134370, Calgary, Alberta
  - GI Research & Associates /ID# 132169, Edmonton, Alberta
  - LAIR Centre /ID# 130970, Vancouver, British Columbia
  - Vancouver Infectious Diseases Centre /ID# 134369, Vancouver, British Columbia
  - GIRI Gastrointestinal Research Institute /ID# 132171, Vancouver, British Columbia
  - University of Manitoba / Health Scuience Centre / John Buhler Research Centre /ID# 130969, Winnipeg, Manitoba
  - Saint John Regional Hospital /ID# 131210, Saint John, New Brunswick
  - Ottawa Hospital Research Institute /ID# 132170, Ottawa, Ontario
  - Toronto General Hospital /ID# 132134, Toronto, Ontario
  - Toronto Liver Centre /ID# 132168, Toronto, Ontario
  - Toronto Digestive Disease Asso /ID# 130968, Vaughan, Ontario
  - Clinique Medicale L'Actuel /ID# 132167, Montreal, Quebec
  - Jewish General Hospital /ID# 132165, Montreal, Quebec
  - Royal Victoria Hospital / McGill University Health Centre /ID# 132166, Montreal, Quebec
  - CHU de Quebec-Université Laval hôpital CHUL /ID# 132132, Québec, Quebec
- Denmark (3):
  - Kobenhavns Universitet - Hvidovre Hospital (HH) /ID# 131031, Hvidovre, Capital Region
  - Odense University Hospital /ID# 131029, Odense C, Region Syddanmark
  - Aarhus Univ Hospital, Skejby /ID# 131030, Aarhus
- Finland (2):
  - Helsinki University Hospital /ID# 131034, Helsinki, Uusimaa
  - Turku University Hospital /ID# 131032, Turku
- France (12):
  - Hopital Saint Joseph /ID# 132177, Marseille, Bouches-du-Rhone
  - CHU Limoges - Dupuytren 1 /ID# 131038, Limoges, Franche-Comte
  - Hopital Haut-Lévêque /ID# 131036, Pessac, Gironde
  - Hopital Saint Eloi /ID# 131037, Montpellier, Herault
  - CHU de Nantes, Hotel Dieu -HME /ID# 132179, Nantes, Pays de la Loire Region
  - Hopital Jean Verdier /ID# 135877, Bondy
  - CHU Grenoble - Hopital Michallon /ID# 131041, La Tronche
  - HCL - Hopital de la Croix-Rousse /ID# 131042, Lyon
  - Duplicate_Hopital lArchet 2 /ID# 131040, Nice
  - CHRU Pontchaillou /ID# 132173, Rennes
  - CHU Strasbourg - Hopital Civil /ID# 132174, Strasbourg
  - Hopital Universitaire Purpan Hopital Rangueil /ID# 131035, Toulouse
- Germany (12):
  - Universitaetsklinikum Freiburg /ID# 131044, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitaetsklinik Heidelberg /ID# 134371, Heidelberg, Baden-Wurttemberg
  - Universitaetsklinikum Tuebingen Medizinische Klinik /ID# 131045, Tübingen, Baden-Wurttemberg
  - LMU Klinikum der Universitat Muchen /ID# 131049, Munich, Bavaria
  - Universitaetsklinikum Frankfurt /ID# 131055, Frankfurt am Main, Hesse
  - Zentru fur HIV und Heaptogastroenterologie /ID# 131052, Düsseldorf, North Rhine-Westphalia
  - Gastroenterologische Gemeinschaftspraxis Herne /ID# 131050, Herne, North Rhine-Westphalia
  - Medizinische Klinik mit Schwerpunkt Hepatologie und Gastroenterologie /ID# 131053, Berlin
  - Universitaetsklinikum Essen /ID# 131048, Essen
  - Universitaetsklinikum Hamburg-Eppendorf (UKE) /ID# 131051, Hamburg
  - Medizinische Hochschule Hannover /ID# 131054, Hanover
  - Centrum für interdisziplinaere Medizin /ID# 131046, Münster
- Greece (3):
  - General Hospital of Athens Ippokratio /ID# 131057, Athens, Attica
  - General Hospital of Athens Laiko /ID# 131088, Athens, Attica
  - General University Hospital of Alexandroupolis /ID# 131056, Alexandroupoli
- Ireland (3):
  - Beaumont Hospital /ID# 131089, Beaumont, Dublin
  - St James Hospital /ID# 132180, Dublin, Dublin
  - St Vincent's University Hospital /ID# 132181, Elm Park, Dublin
- Israel (4):
  - The Chaim Sheba Medical Center /ID# 131092, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 132182, Tel Aviv, Tel Aviv
  - Rambam Health Care Campus /ID# 131090, Haifa
  - The Lady Davis Carmel Medical Center /ID# 131091, Haifa
- Italy (22):
  - Duplicate_A.O.U. Policlinico S.Orsola-Malpighi /ID# 131095, Bologna, Emilia-Romagna
  - Azienda Ospedaliero-Universitaria di Ferrara-Arcispedale Sant Anna /ID# 131102, Cona, Ferrara
  - Fondazione di Religione e di Culto Casa Sollievo della Sofferenza /ID# 132190, San Giovanni Rotondo, Foggia
  - Policlinico Agostino Gemelli /ID# 131098, Rome, Lazio
  - Ospedale San Raffaele IRCCS /ID# 131093, Milan, Lombardy
  - Fondazione PTV Policlinico Tor Vergata /ID# 132185, Rome, Roma
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII (Presidio Papa Giovanni /ID# 132188, Bergamo
  - Azienda Ospedaliero Universitaria Careggi /ID# 132197, Florence
  - Azienda Ospedaliera Universitaria Ospedali Riuniti /ID# 132195, Foggia
  - A.O.U. Policlinico G. Martino /ID# 132193, Messina
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico /ID# 131097, Milan
  - Ospedale S Giuseppe /ID# 132194, Milan
  - ASST Santi Paolo e Carlo/Presidio Ospedale San Paolo /ID# 132198, Milan
  - ASST Fatebenefratelli Sacco-Ospedale Sacco /ID# 134372, Milan
  - Azienda Ospedaliera Niguarda Ca' Granda Hospital /ID# 131104, Milan
  - Azienda Ospedaliera Universitaria Federico II /ID# 131096, Napoli
  - Azienda Ospedaliera Universitaria Federico II /ID# 132191, Napoli
  - Azienda Ospedaliera Universitaria Paolo Giaccone /ID# 132184, Palermo
  - Azienda Ospedaliero-Universitaria di Parma /ID# 132183, Parma
  - Azienda Ospedaliera Universitaria "San Giovanni di Dio e Ruggi d'Aragona /ID# 132192, Salerno
  - A.O.U. Citta della Salute e della Scienza di Torino /ID# 131100, Turin
  - Azienda Ospedaliera Universitaria Friuli Centrale/Presidio Ospedaliero Universit /ID# 132196, Udine
- Mexico (6):
  - Hospital General de Tijuana /ID# 130972, Tijuana, Estado de Baja California
  - Cife /Id# 130974, Guadalajara, Jalisco
  - Instituto Nacional de Clencias Medicas y Nutricion Salvador Zubrian Departament /ID# 130975, Distrito Federal
  - CIF-BIOTEC/Medica Sur /ID# 134971, Mexico City
  - ITESM campus Ciudad de Mexico /ID# 132383, Mexico City
  - Instituto Metropolitano de Inv /ID# 132201, Tlalpan
- Netherlands (3):
  - Erasmus Medisch Centrum /ID# 132206, Rotterdam, South Holland
  - Academisch Medisch Centrum /ID# 132205, Amsterdam
  - Leids Universitair Medisch Centrum /ID# 132204, Leiden
- Norway (3):
  - Akershus Universitetssykehus_MAIN /ID# 132212, Lorenskog, Akershus
  - St. Olavs Hospital HF /ID# 132213, Trondheim, Sor-Trondelag
  - Stavanger University Hospital /ID# 132211, Stavanger
- Poland (6):
  - Wojewodzki Szpital Obserwacyjno-Zakazny im. Tadeusza Browicza /ID# 131106, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 w Lublinie /ID# 131115, Lublin, Lublin Voivodeship
  - Wojewodzki Szpital Zakazny /ID# 131112, Warsaw, Masovian Voivodeship
  - Uniwersytecki Szpital Kliniczny w Bialymstoku /ID# 131108, Bialystok, Podlaskie Voivodeship
  - ID Clinic /ID# 131111, Mysłowice, Silesian Voivodeship
  - Wojewodzki Specjalistyczny Szpital im. dr. W. Bieganskiego /ID# 131107, Lodz, Łódź Voivodeship
- Portugal (4):
  - Centro Hospitalar e Universitario de Coimbra, EPE /ID# 131119, Coimbra
  - Centro Hospitalar Universitario Lisboa Central, EPE - Hospital dos Capuchos /ID# 131116, Lisbon
  - Centro Hospitalar Universitário de Lisboa Norte, EPE - Hospital de Santa Maria /ID# 131118, Lisbon
  - Centro Hospitalar Universitário do Porto, EPE - Hospital Santo António /ID# 131117, Porto
- Romania (5):
  - Duplicate_Institutul National de Boli Infectioase Prof. Dr. Matei Bals /ID# 131120, Sector 2, București
  - Institutul Clinic Fundeni /ID# 131121, Sector 2, București
  - Spitalul Clinic de Boli Infectioase Si Pneumoftiziologie Dr. Victor Babes /Id# 131126, Timișoara, Timiș County
  - Institutul Nat. de Boli Infectioase /ID# 131124, Bucharest
  - SC Gastromedica SRL /ID# 131127, Iași
- Russia (16):
  - Medical Company Hepatolog /ID# 132277, Samara, Samara Oblast
  - Republican Clinical Infectious Diseases Hospital n.a. Professor A. F. Agafonov /ID# 132270, Kazan', Tatarstan, Respublika
  - South-Ural State Med. Academy /ID# 132274, Chelyabinsk
  - Kuzbass Center for Prevention and Fight agains AIDS /ID# 132269, Kemerovo
  - Krasnoyarsk Regional Center for the Prevention and Control of AIDS /ID# 132278, Krasnoyarsk
  - Moscow Clinical Scientific Center n.a. Loginov /ID# 132266, Moscow
  - Central Clinical Hospital of Russian Academy of Science /ID# 132289, Moscow
  - I. M. Sechenov First Moscow State Medical University /ID# 132275, Moscow
  - City Clinical Hospital #24 /ID# 132268, Moscow
  - Research Institute of Emergency Medicine named after V.I. N.V. Sklifosovsky /ID# 132288, Moscow
  - Clinical Infectious Diseases Hospital #1 /ID# 132272, Novosibirsk
  - Samara State Medical University /ID# 136913, Samara
  - Stavropol State Medical University /ID# 132279, Stavropol
  - Tolyatti City Clinical Hospital #1 /ID# 132273, Tolyatti
  - Multidisciplinary Consultative and Diagnostic Center /ID# 131130, Tyumen
  - Sverdlovsk Regional Clinical Hospital #1 /ID# 132267, Yekaterinburg
- Saudi Arabia (3):
  - King Abdulaziz Medical City /ID# 145129, Jeddah
  - Ministry Nat Guard Hosp Health /ID# 145126, Riyadh
  - King Khalid University Hospita /ID# 132291, Riyadh
- Spain (15):
  - Hospital Universitari Son Espases /ID# 131140, Palma de Mallorca, Balearic Islands
  - Hospital Universitario Germans Trias i Pujol /ID# 132293, Badalona, Barcelona
  - Hospital Unversitario Marques de Valdecilla /ID# 131141, Santander, Cantabria
  - Hospital Donostia /ID# 131144, Donostia / San Sebastian, Guipuzcoa
  - Hospital General Universitario Santa Lucia /ID# 131139, Cartagena, Murcia
  - Hospital Universitario Central de Asturias /ID# 131138, Oviedo, Principality of Asturias
  - OSI Ezkerraldea-Enkarterri-Cruces /ID# 131143, Barakaldo, Vizcaya
  - Hospital Universitario A Coruna - CHUAC /ID# 131137, A Coruña
  - Hospital Universitario Reina Sofia /ID# 131135, Córdoba
  - Hospital Universitario de la Princesa /ID# 131131, Madrid
  - Hospital Universitario 12 de Octubre /ID# 131133, Madrid
  - Hospital Universitario La Paz /ID# 131132, Madrid
  - Hospital Universitario Virgen de la Victoria /ID# 131136, Málaga
  - Hospital Universitario Virgen del Rocio /ID# 131134, Seville
  - Hospital Clinico Universitario Lozano Blesa /ID# 132292, Zaragoza
- Sweden (3):
  - Skane University hospital /ID# 131146, Malmo, Skåne County
  - Karolinska University Hospital Solna /ID# 131145, Solna, Stockholm County
  - Sahlgrenska University Hospital /ID# 131147, Gothenburg, Västra Götaland County
- Switzerland (3):
  - Kantonsspital St. Gallen /ID# 131148, Sankt Gallen, Canton of St. Gallen
  - Universitätsspital Zürich /ID# 134881, Zurich, Canton of Zurich
  - Inselspital, Universitätsspital Bern /ID# 132294, Bern
- Turkey (Türkiye) (7):
  - Izmir Tepecik Training and Research Hospital /ID# 134968, Konak, İzmir
  - Hacettepe University Faculty of Medicine /ID# 131150, Ankara
  - Ankara Univ Medical Faculty /ID# 131151, Ankara
  - Uludag University Medical Faculty /ID# 132297, Bursa
  - Istanbul University Istanbul Medical Faculty /ID# 131153, Istanbul
  - Ege University Medical Faculty /ID# 132298, Izmir
  - Karadeniz University /ID# 131152, Trabzon
- United Kingdom (15):
  - Duplicate_University Hospitals Dorset NHS Foundation Trust /ID# 132306, Poole, Dorset
  - University Hospital Southampton NHS Foundation Trust /ID# 131161, Southampton, Hampshire
  - Barts Health NHS Trust /ID# 132302, London, London, City of
  - The Royal Free London NHS Foundation Trust /ID# 131159, London, London, City of
  - Duplicate_Nottingham University Nottingham University Hospitals NHS Trust /ID# 131155, Nottingham, Nottinghamshire
  - NHS Greater Glasgow and Clyde /ID# 131162, Glasgow, Scotland
  - University Hospitals Birmingham NHS Foundation Trust /ID# 131154, Birmingham
  - Duplicate_NHS Tayside /ID# 132300, Dundee
  - NHS Lothian /ID# 134368, Edinburgh
  - Leeds Teaching Hospitals NHS Trust /ID# 132305, Leeds
  - King's College Hospital NHS Foundation Trusts /ID# 131157, London
  - University Hospital Plymouth NHS Trust /ID# 131160, Plymouth
  - Portsmouth Hospitals University NHS Trust /ID# 131158, Portsmouth
  - Northern Care Alliance NHS Group /ID# 131156, Salford
  - St George's University Hospitals NHS Foundation Trust /ID# 132301, Tooting

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing, please refer to the link below.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Use Agreement (DUA). For more information on the process, or to submit a request, visit the following link.
URL: https://vivli.org/ourmember/abbvie/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Safety population: All participants enrolled in this study (M14-423; TOPAZ-I) who received at least one dose of study drug
Period: Overall Study
Arm/Group | ABT-450/r/ABT-267 Plus ABT-333 With or Without Ribavirin (RBV)
Started | 1596
Completed | 1258
Not Completed | 338
Not completed — Adverse Event | 24
Not completed — Withdrew consent | 96
Not completed — Lost to Follow-up | 126
Not completed — COVID-19 infection | 2
Not completed — COVID-19 logistical restrictions | 33
Not completed — Other, not specified | 57

BASELINE CHARACTERISTICS:
Population: Safety population: All participants enrolled in this study (M14-423; TOPAZ-I) who received at least one dose of study drug
Arm/Group | ABT-450/r/ABT-267 Plus ABT-333 With or Without Ribavirin (RBV)
Number analyzed (Participants) | 1596
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (11.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 800
  Male | 796
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 1544
  Black or African American | 10
  Asian | 39
  American Indian or Alaska Native | 1
  Native Hawaiian or Other Pacific Islander | 0
  Multiple | 2
HCV Genotype 1 Subtype [Count of Participants; unit: Participants]
  GT1b without cirrhosis | 757
  GT1b with compensated cirrhosis | 142
  GT1 Non-b without cirrhosis | 597
  GT1 Non-b with compensated cirrhosis | 97
  Missing | 3
Prior HCV Treatment History [Count of Participants; unit: Participants]
  Treatment Naïve | 782
  Treatment Experienced | 814

OUTCOME MEASURES:

1. Primary Outcome: All-Cause Death: Time to Event
Description: Time to all-cause death was defined as the number of days from the first day of study drug dosing for the participant to the date of death. All deaths were to be included, regardless of whether the death occurred while the participant was still taking study drug or had previously discontinued study drug. If the participant did not die, their data was to be censored at the date of their last available assessment of clinical outcomes. For participants with no post-baseline assessment, the participant's data was to be censored on the first day of study drug dosing. The event-free survival rates were estimated using Kaplan-Meier methodology and incidence estimates are presented with 95% confidence intervals. The pre-specified analysis of all-cause death included pooled data from TOPAZ-I (this study) and the companion study TOPAZ-II (M14-222; NCT02167945).
Time Frame: At Post-Treatment Weeks 52, 104, 156, 208, and 260
Population: Intent-to-treat (ITT) population: all enrolled participants in this study (TOPAZ-I; M14-423; ITT-I) and in companion study M14-422 (TOPAZ-II; NCT02167945; ITT-II) who received at least one dose of study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Participants in Studies M14-222 and M14-423 Who Did Not Achieve SVR12; Participants in Studies M14-222 and M14-423 Who Achieved SVR12: SVR12 was defined as hepatitis C virus ribonucleic acid (HCV RNA) less than the lower limit of quantification (LLOQ) 12 weeks after the last actual dose of study drug.
Arm/Group | Participants in Studies M14-222 and M14-423 Who Did Not Achieve SVR12 | Participants in Studies M14-222 and M14-423 Who Achieved SVR12
Number analyzed (Participants) | 77 | 2134
percentage of participants
  Kaplan-Meier estimate at PT Week 52 | 8.3 [3.1 to 21.2] | 0.1 [0.1 to 0.4]
  Kaplan-Meier estimate at PT Week 104 | 8.3 [3.1 to 21.2] | 0.7 [0.4 to 1.1]
  Kaplan-Meier estimate at PT Week 156 | 8.3 [3.1 to 21.2] | 1.2 [0.8 to 1.8]
  Kaplan-Meier estimate at PT Week 208 | 8.3 [3.1 to 21.2] | 1.5 [1.1 to 2.2]
  Kaplan-Meier estimate at PT Week 260 | 8.3 [3.1 to 21.2] | 2.0 [1.5 to 2.8]
Statistical Analysis 1: Comparison: Participants in Studies M14-222 and M14-423 Who Did Not Achieve SVR12 vs Participants in Studies M14-222 and M14-423 Who Achieved SVR12; Comparisons between participants in studies M14-222 and M14-423 who achieved SVR12 and those who did not were performed using a log-rank test; Test type: Superiority; p < 0.001, Log-rank test
Statistical Analysis 2: Comparison: Participants in Studies M14-222 and M14-423 Who Did Not Achieve SVR12 vs Participants in Studies M14-222 and M14-423 Who Achieved SVR12; A Cox proportional hazards (PH) model was constructed. The covariates for the model included baseline age, BMI, HCV genotype 1 subtype (1b, non-1b), IL28B genotype (CC, non-CC), prior treatment history (naive, experienced), baseline HCV RNA levels, baseline fibrosis stage (F0-1, F2, F3, F4), baseline albumin, baseline creatinine clearance, baseline platelet count, history of diabetes (yes, no), APRI, race (white, other), and alcohol use status (current, former, non-drinker); Test type: Superiority; p < 0.001, Cox proportional hazards model; Cox Proportional Hazard Ratio = 0.126, 95% CI 2-sided [0.044 to 0.358] — The estimated value represents the hazard ratio for developing the event in the group of participants in studies M14-222 and M14-423 who achieved SVR12 compared to the group of participants in studies M14-222 and M14-423 who didn't achieve SVR12

2. Primary Outcome: Liver-Related Death: Time to Event
Description: Time to liver-related death was defined as days from the 1st day of study drug dosing for the subject to date of liver-related death. All liver-related deaths were to be included, regardless of whether the death occurred while subject was still taking study drug or had previously discontinued study drug. If the subject didn't experience event of interest nor had died (all-cause death), their data was to be censored at date of last available assessment. For those with no post-baseline assessment, data was to be censored on 1st day of study drug dosing. All-cause death was a censoring event for liver-related death. The event-free survival rates were estimated using Kaplan-Meier methodology and incidence estimates are presented with 95% confidence intervals. The pre-specified analysis of liver-related death included pooled data from TOPAZ-I (this study) and the companion study TOPAZ-II (M14-222; NCT02167945).
Time Frame: At Post-Treatment Weeks 52, 104, 156, 208, and 260
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants in Studies M14-222 and M14-423 Who Did Not Achieve SVR12 | Participants in Studies M14-222 and M14-423 Who Achieved SVR12
Number analyzed (Participants) | 77 | 2134
percentage of participants
  Kaplan-Meier estimate at PT Week 52 | 1.4 [0.2 to 9.6] | 0 [NA to NA] — Confidence interval is not calculable due to zero events at this visit
  Kaplan-Meier estimate at PT Week 104 | 1.4 [0.2 to 9.6] | 0 [NA to NA] — Confidence interval is not calculable due to zero events at this visit
  Kaplan-Meier estimate at PT Week 156 | 1.4 [0.2 to 9.6] | 0.1 [0.1 to 0.4]
  Kaplan-Meier estimate at PT Week 208 | 1.4 [0.2 to 9.6] | 0.1 [0.1 to 0.4]
  Kaplan-Meier estimate at PT Week 260 | 1.4 [0.2 to 9.6] | 0.1 [0.1 to 0.4]
Statistical Analysis 1: Comparison: Participants in Studies M14-222 and M14-423 Who Did Not Achieve SVR12 vs Participants in Studies M14-222 and M14-423 Who Achieved SVR12; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Log-rank test
Statistical Analysis 2: Comparison: Participants in Studies M14-222 and M14-423 Who Did Not Achieve SVR12 vs Participants in Studies M14-222 and M14-423 Who Achieved SVR12; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.007, Cox proportional hazards model; Cox Proportional Hazard Ratio = 0.031, 95% CI 2-sided [0.003 to 0.380] — [estimate comment as in outcome 1, analysis 2]

3. Primary Outcome: Liver Decompensation: Time to Event
Description: Time to liver decompensation was defined as number of days from the 1st day of study drug dosing for the participant to the date of liver decompensation. All liver decompensation was to be included, regardless of whether it occurred while the participant was still taking study drug or had previously discontinued study drug. If the participant didn't experience the event of interest nor had died (all-cause death), their data was to be censored at the date of their last available assessment of clinical outcomes. For participants with no post-baseline assessment, their data was to be censored on the 1st day of study drug dosing. All-cause death was a censoring event for liver decompensation. The event-free survival rates were estimated using Kaplan-Meier methodology and incidence estimates are presented with 95% confidence intervals. The pre-specified analysis of liver decompensation included pooled data from TOPAZ-I (this study) and the companion study TOPAZ-II (M14-222; NCT02167945).
Time Frame: At Post-Treatment Weeks 52, 104, 156, 208, and 260
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants in Studies M14-222 and M14-423 Who Did Not Achieve SVR12 | Participants in Studies M14-222 and M14-423 Who Achieved SVR12
Number analyzed (Participants) | 77 | 2134
percentage of participants
  Kaplan-Meier estimate at PT Week 52 | 4.5 [1.5 to 13.4] | 0.2 [0.1 to 0.5]
  Kaplan-Meier estimate at PT Week 104 | 4.5 [1.5 to 13.4] | 0.2 [0.1 to 0.5]
  Kaplan-Meier estimate at PT Week 156 | 4.5 [1.5 to 13.4] | 0.3 [0.1 to 0.6]
  Kaplan-Meier estimate at PT Week 208 | 4.5 [1.5 to 13.4] | 0.3 [0.2 to 0.7]
  Kaplan-Meier estimate at PT Week 260 | 4.5 [1.5 to 13.4] | 0.5 [0.2 to 0.9]
Statistical Analysis 1: Comparison: Participants in Studies M14-222 and M14-423 Who Did Not Achieve SVR12 vs Participants in Studies M14-222 and M14-423 Who Achieved SVR12; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Log-rank test
Statistical Analysis 2: Comparison: Participants in Studies M14-222 and M14-423 Who Did Not Achieve SVR12 vs Participants in Studies M14-222 and M14-423 Who Achieved SVR12; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.001, Cox proportional hazards model; Cox Proportional Hazard Ratio = 0.038, 95% CI 2-sided [0.009 to 0.156] — [estimate comment as in outcome 1, analysis 2]

4. Primary Outcome: Liver Transplantation: Time to Event
Description: Time to liver transplantation was defined as days from 1st day of study drug dosing for subject to date of liver transplantation. All liver transplantation was to be included, whether it occurred while the subject was still taking study drug or had previously discontinued study drug. If the subject didn't experience event of interest nor had died (all-cause death), their data was to be censored at the date of their last available assessment. For those with no post-baseline assessment, data was to be censored on 1st day of study drug dosing. All-cause death was a censoring event for liver transplantation. The event-free survival rates were estimated using Kaplan-Meier methodology and incidence estimates are presented with 95% confidence intervals. The pre-specified analysis of liver transplantation included pooled data from TOPAZ-I (this study) and the companion study TOPAZ-II (M14-222; NCT02167945).
Time Frame: At Post-Treatment Weeks 52, 104, 156, 208, and 260
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants in Studies M14-222 and M14-423 Who Did Not Achieve SVR12 | Participants in Studies M14-222 and M14-423 Who Achieved SVR12
Number analyzed (Participants) | 77 | 2134
percentage of participants
  Kaplan-Meier estimate at PT Week 52 | 0 [NA to NA] — Confidence interval is not calculable due to zero events at this visit | 0 [NA to NA] — Confidence interval is not calculable due to zero events at this visit
  Kaplan-Meier estimate at PT Week 104 | 0 [NA to NA] — Confidence interval is not calculable due to zero events at this visit | 0 [NA to NA] — Confidence interval is not calculable due to zero events at this visit
  Kaplan-Meier estimate at PT Week 156 | 0 [NA to NA] — Confidence interval is not calculable due to zero events at this visit | 0.1 [0.1 to 0.4]
  Kaplan-Meier estimate at PT Week 208 | 0 [NA to NA] — Confidence interval is not calculable due to zero events at this visit | 0.1 [0.1 to 0.4]
  Kaplan-Meier estimate at PT Week 260 | 0 [NA to NA] — Confidence interval is not calculable due to zero events at this visit | 0.2 [0.1 to 0.5]
Statistical Analysis 1: Comparison: Participants in Studies M14-222 and M14-423 Who Did Not Achieve SVR12 vs Participants in Studies M14-222 and M14-423 Who Achieved SVR12; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.860, Log-rank test
Statistical Analysis 2: Comparison: Participants in Studies M14-222 and M14-423 Who Did Not Achieve SVR12 vs Participants in Studies M14-222 and M14-423 Who Achieved SVR12; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.997, Cox proportional hazards model — The Hazard Ratio for experiencing the event in the group of participants in studies M14-222 and M14-423 who achieved SVR12 compared to those who did not achieve SVR12 is infinite and the CI is not bounded due to zero events in one of the groups

5. Primary Outcome: Hepatocellular Carcinoma: Time to Event
Description: Time to hepatocellular carcinoma (HCC) was defined as number of days from 1st day of study drug dosing for subject to date of hepatocellular carcinoma. All HCC was to be included, whether it occurred while subject was still taking study drug or had previously discontinued study drug. If the subject didn't experience the event of interest nor had died (all-cause death), their data was to be censored at the date of their last available assessment. For those with no post-baseline assessment, their data was to be censored on the 1st day of study drug dosing. All-cause death was a censoring event for HCC. The event-free survival rates were estimated using Kaplan-Meier methodology and incidence estimates are presented with 95% confidence intervals. The pre-specified analysis of hepatocellular carcinoma included pooled data from TOPAZ-I (this study) and the companion study TOPAZ-II (M14-222; NCT02167945).
Time Frame: At Post-Treatment Weeks 52, 104, 156, 208, and 260
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants in Studies M14-222 and M14-423 Who Did Not Achieve SVR12 | Participants in Studies M14-222 and M14-423 Who Achieved SVR12
Number analyzed (Participants) | 77 | 2134
percentage of participants
  Kaplan-Meier estimate at PT Week 52 | 0 [NA to NA] — Confidence interval is not calculable due to zero events at this visit | 0.2 [0.1 to 0.5]
  Kaplan-Meier estimate at PT Week 104 | 0 [NA to NA] — Confidence interval is not calculable due to zero events at this visit | 0.4 [0.2 to 0.8]
  Kaplan-Meier estimate at PT Week 156 | 0 [NA to NA] — Confidence interval is not calculable due to zero events at this visit | 0.5 [0.3 to 1.0]
  Kaplan-Meier estimate at PT Week 208 | 0 [NA to NA] — Confidence interval is not calculable due to zero events at this visit | 0.6 [0.4 to 1.1]
  Kaplan-Meier estimate at PT Week 260 | 0 [NA to NA] — Confidence interval is not calculable due to zero events at this visit | 0.9 [0.5 to 1.4]
Statistical Analysis 1: Comparison: Participants in Studies M14-222 and M14-423 Who Did Not Achieve SVR12 vs Participants in Studies M14-222 and M14-423 Who Achieved SVR12; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.608, Log-rank test
Statistical Analysis 2: Comparison: Participants in Studies M14-222 and M14-423 Who Did Not Achieve SVR12 vs Participants in Studies M14-222 and M14-423 Who Achieved SVR12; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.992, Cox proportional hazards model — [p-value comment as in outcome 4, analysis 2]

6. Primary Outcome: All-Cause Death, Liver-Related Death, Liver Decompensation, Liver Transplantation, Hepatocellular Carcinoma: Time to Event
Description: Time to the composite of clinical outcomes is the time to the first occurrence of all-cause death, liver-related death, liver decompensation, liver transplantation, or hepatocellular carcinoma. All first occurrences were to be included, regardless of whether it occurred while the participant was still taking study drug or had previously discontinued study drug. If the participant did not experience any of these events, their data was to be censored at the date of their last available assessment of clinical outcomes. For participants with no post-baseline assessment, the participant's data was to be censored on the first day of study drug dosing. The event-free survival rates were estimated using Kaplan-Meier methodology and incidence estimates are presented with 95% confidence intervals. Pre-specified analysis included pooled data from this study and from TOPAZ-II; NCT02167945.
Time Frame: At Post-Treatment Weeks 52, 104, 156, 208, and 260
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants in Studies M14-222 and M14-423 Who Did Not Achieve SVR12 | Participants in Studies M14-222 and M14-423 Who Achieved SVR12
Number analyzed (Participants) | 77 | 2134
percentage of participants
  Kaplan-Meier estimate at PT Week 52 | 11.4 [5.2 to 24.2] | 0.5 [0.3 to 0.9]
  Kaplan-Meier estimate at PT Week 104 | 11.4 [5.2 to 24.2] | 1.2 [0.8 to 1.8]
  Kaplan-Meier estimate at PT Week 156 | 11.4 [5.2 to 24.2] | 1.9 [1.4 to 2.6]
  Kaplan-Meier estimate at PT Week 208 | 11.4 [5.2 to 24.2] | 2.3 [1.7 to 3.1]
  Kaplan-Meier estimate at PT Week 260 | 11.4 [5.2 to 24.2] | 3.2 [2.5 to 4.1]
Statistical Analysis 1: Comparison: Participants in Studies M14-222 and M14-423 Who Did Not Achieve SVR12 vs Participants in Studies M14-222 and M14-423 Who Achieved SVR12; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Log-rank test
Statistical Analysis 2: Comparison: Participants in Studies M14-222 and M14-423 Who Did Not Achieve SVR12 vs Participants in Studies M14-222 and M14-423 Who Achieved SVR12; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.001, Cox proportional hazards model; Cox Proportional Hazard Ratio = 0.133, 95% CI 2-sided [0.057 to 0.313] — [estimate comment as in outcome 1, analysis 2]

7. Secondary Outcome: Change From Baseline in FibroScan Score by SVR12 Status
Description: The FibroScan test is a validated non-invasive test used to assess liver fibrosis in participants with chronic liver disease, and it was performed at study sites where it was available. For participants with Hepatitis C infection, a FibroScan score of 2-7 kPa indicates no liver scarring or mild scarring; a score of 8 or 9 is associated with moderate liver scarring; 9-14 indicates severe liver scarring; and 14 or higher is indicative of advanced liver scarring, cirrhosis. Negative changes from baseline indicate improvement in liver fibrosis.
Time Frame: At the final treatment visit and Post-Treatment Weeks 12, 24, 52, 104, 156, 208, and 260
Population: ITT-I population: all participants enrolled in this study (M14-423; TOPAZ-I) who received at least one dose of study drug with available data
Measure: Mean (Standard Deviation); unit: kPa
Groups:
- Participants in Study M14-423 Who Did Not Achieve SVR12; Participants in Study M14-423 Who Achieved SVR12: SVR12 was defined as hepatitis C virus ribonucleic acid (HCV RNA) less than the lower limit of quantification (LLOQ) 12 weeks after the last actual dose of study drug.
Arm/Group | Participants in Study M14-423 Who Did Not Achieve SVR12 | Participants in Study M14-423 Who Achieved SVR12
Number analyzed (Participants) | 22 | 1187
kPa
  At the final treatment visit: number analyzed (Participants) | 22 | 1015
  At the final treatment visit | -2.55 (3.282) | -1.41 (4.283)
  Post-Treatment Week 12: number analyzed (Participants) | 18 | 1171
  Post-Treatment Week 12 | -1.81 (2.624) | -1.76 (4.213)
  Post-Treatment Week 24: number analyzed (Participants) | 18 | 1175
  Post-Treatment Week 24 | -1.26 (3.211) | -1.98 (4.363)
  Post-Treatment Week 52: number analyzed (Participants) | 13 | 1187
  Post-Treatment Week 52 | -0.30 (1.986) | -2.46 (4.858)
  Post-Treatment Week 104: number analyzed (Participants) | 13 | 1122
  Post-Treatment Week 104 | -0.35 (3.306) | -2.80 (5.195)
  Post-Treatment Week 156: number analyzed (Participants) | 12 | 1073
  Post-Treatment Week 156 | -0.37 (3.999) | -2.92 (5.249)
  Post-Treatment Week 208: number analyzed (Participants) | 12 | 978
  Post-Treatment Week 208 | -0.88 (2.445) | -3.08 (5.560)
  Post-Treatment Week 260: number analyzed (Participants) | 9 | 860
  Post-Treatment Week 260 | -1.31 (3.706) | -3.08 (5.662)
Statistical Analysis 1: Comparison: Participants in Study M14-423 Who Did Not Achieve SVR12 vs Participants in Study M14-423 Who Achieved SVR12; Final Treatment Visit The effect of sustained virologic response on change from baseline in FibroScan score was evaluated by comparing mean change from baseline between subjects who achieved SVR12 and those who did not using ANCOVA analyses. SVR12 status was included as a factor and baseline FibroScan score was included as a covariate in the ANCOVA model; Test type: Superiority; p = 0.151, ANCOVA; LS Mean Difference = 1, 95% CI 2-sided [-0.37 to 2.37], Standard Error of Mean 0.7 — Difference = with SVR12 minus without SVR12
Statistical Analysis 2: Comparison: Participants in Study M14-423 Who Did Not Achieve SVR12 vs Participants in Study M14-423 Who Achieved SVR12; Post-Treatment Week 12 The effect of sustained virologic response on change from baseline in FibroScan score was evaluated by comparing mean change from baseline between subjects who achieved SVR12 and those who did not using ANCOVA analyses. SVR12 status was included as a factor and baseline FibroScan score was included as a covariate in the ANCOVA model; Test type: Superiority; p = 0.878, ANCOVA; LS Mean Difference = -0.12, 95% CI 2-sided [-1.64 to 1.4], Standard Error of Mean 0.78 — Difference = with SVR12 minus without SVR12
Statistical Analysis 3: Comparison: Participants in Study M14-423 Who Did Not Achieve SVR12 vs Participants in Study M14-423 Who Achieved SVR12; Post-Treatment Week 24 The effect of sustained virologic response on change from baseline in FibroScan score was evaluated by comparing mean change from baseline between subjects who achieved SVR12 and those who did not using ANCOVA analyses. SVR12 status was included as a factor and baseline FibroScan score was included as a covariate in the ANCOVA model; Test type: Superiority; p = 0.199, ANCOVA; LS Mean Difference = -0.92, 95% CI 2-sided [-2.33 to 0.48], Standard Error of Mean 0.72 — Difference = with SVR12 minus without SVR12
Statistical Analysis 4: Comparison: Participants in Study M14-423 Who Did Not Achieve SVR12 vs Participants in Study M14-423 Who Achieved SVR12; Post-Treatment Week 52 The effect of sustained virologic response on change from baseline in FibroScan score was evaluated by comparing mean change from baseline between subjects who achieved SVR12 and those who did not using ANCOVA analyses. SVR12 status was included as a factor and baseline FibroScan score was included as a covariate in the ANCOVA model; Test type: Superiority; p = 0.021, ANCOVA; LS Mean Difference = -2.16, 95% CI 2-sided [-4 to -0.33], Standard Error of Mean 0.93 — Difference = with SVR12 minus without SVR12
Statistical Analysis 5: Comparison: Participants in Study M14-423 Who Did Not Achieve SVR12 vs Participants in Study M14-423 Who Achieved SVR12; Post-Treatment Week 104 The effect of sustained virologic response on change from baseline in FibroScan score was evaluated by comparing mean change from baseline between subjects who achieved SVR12 and those who did not using ANCOVA analyses. SVR12 status was included as a factor and baseline FibroScan score was included as a covariate in the ANCOVA model; Test type: Superiority; p = 0.006, ANCOVA; LS Mean Difference = -2.47, 95% CI 2-sided [-4.22 to -0.71], Standard Error of Mean 0.89 — Difference = with SVR12 minus without SVR12
Statistical Analysis 6: Comparison: Participants in Study M14-423 Who Did Not Achieve SVR12 vs Participants in Study M14-423 Who Achieved SVR12; Post-Treatment Week 156 The effect of sustained virologic response on change from baseline in FibroScan score was evaluated by comparing mean change from baseline between subjects who achieved SVR12 and those who did not using ANCOVA analyses. SVR12 status was included as a factor and baseline FibroScan score was included as a covariate in the ANCOVA model; Test type: Superiority; p = 0.005, ANCOVA; LS Mean Difference = -2.58, 95% CI 2-sided [-4.38 to -0.79], Standard Error of Mean 0.92 — Difference = with SVR12 minus without SVR12
Statistical Analysis 7: Comparison: Participants in Study M14-423 Who Did Not Achieve SVR12 vs Participants in Study M14-423 Who Achieved SVR12; Post-Treatment Week 208 The effect of sustained virologic response on change from baseline in FibroScan score was evaluated by comparing mean change from baseline between subjects who achieved SVR12 and those who did not using ANCOVA analyses. SVR12 status was included as a factor and baseline FibroScan score was included as a covariate in the ANCOVA model; Test type: Superiority; p = 0.172, ANCOVA; LS Mean Difference = -1.36, 95% CI 2-sided [-3.32 to 0.59], Standard Error of Mean 1 — Difference = with SVR12 minus without SVR12
Statistical Analysis 8: Comparison: Participants in Study M14-423 Who Did Not Achieve SVR12 vs Participants in Study M14-423 Who Achieved SVR12; Post-Treatment Week 260 The effect of sustained virologic response on change from baseline in FibroScan score was evaluated by comparing mean change from baseline between subjects who achieved SVR12 and those who did not using ANCOVA analyses. SVR12 status was included as a factor and baseline FibroScan score was included as a covariate in the ANCOVA model; Test type: Superiority; p = 0.322, ANCOVA; LS Mean Difference = -1.13, 95% CI 2-sided [-3.35 to 1.1], Standard Error of Mean 1.14 — Difference = with SVR12 minus without SVR12

8. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks Post-treatment (SVR12)
Description: SVR12 is defined as hepatitis C virus ribonucleic acid (HCV RNA) less than the lower limit of quantification (LLOQ) 12 weeks after the last actual dose of study drug. Flanking imputation, where applicable, was used to impute missing data. After applying flanking imputation, if there was no value in the window but there was an HCV RNA value from a local laboratory present, then it was to be imputed into the SVR window. Otherwise, participants with missing data were counted as failures.
Time Frame: 12 weeks after the last actual dose of study drug
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABT-450/r/ABT-267 Plus ABT-333 With or Without Ribavirin (RBV)
Number analyzed (Participants) | 1596
percentage of participants | 97.0 [96.0 to 97.7]

ADVERSE EVENTS:
Time Frame: All-cause mortality is reported from enrollment to the end of study, up to five years of follow-up. Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from the first dose of study drug until 30 days after the last study drug administration, up to 203 days. After Post-Treatment Week 4 until the end of the study, only SAE of death was to be collected.
Description: All-cause mortality and adverse events: all participants in this study (M14-423; TOPAZ-I) who received at least one dose of study drug
Arm/Group | ABT-450/r/ABT-267 Plus ABT-333 With or Without Ribavirin (RBV)
All-Cause Mortality (participants affected / at risk) | 28/1596
Serious Adverse Events (participants affected / at risk) | 40/1596
Other Adverse Events (participants affected / at risk) | 805/1596
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABT-450/r/ABT-267 Plus ABT-333 With or Without Ribavirin (RBV) (N=1596)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1)
ANGINA UNSTABLE (Cardiac disorders) | 1 (1)
PALPITATIONS (Cardiac disorders) | 1 (1)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1)
ANAL FISSURE (Gastrointestinal disorders) | 1 (1)
ASCITES (Gastrointestinal disorders) | 1 (1)
COLITIS (Gastrointestinal disorders) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 1 (1)
DENTAL CARIES (Gastrointestinal disorders) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 1 (1)
GASTRIC ULCER (Gastrointestinal disorders) | 1 (1)
OESOPHAGEAL VARICES HAEMORRHAGE (Gastrointestinal disorders) | 1 (1)
VARICES OESOPHAGEAL (Gastrointestinal disorders) | 1 (1)
DRUG INTERACTION (General disorders) | 1 (1)
OEDEMA PERIPHERAL (General disorders) | 1 (1)
HEPATIC FAILURE (Hepatobiliary disorders) | 1 (1)
HEPATORENAL SYNDROME (Hepatobiliary disorders) | 1 (1)
APPENDICITIS (Infections and infestations) | 1 (1)
DERMATITIS INFECTED (Infections and infestations) | 1 (1)
ERYSIPELAS (Infections and infestations) | 1 (1)
INFLUENZA (Infections and infestations) | 1 (1)
PERITONITIS BACTERIAL (Infections and infestations) | 1 (1)
PNEUMONIA (Infections and infestations) | 2 (2)
PYELONEPHRITIS (Infections and infestations) | 1 (1)
HEAD INJURY (Injury, poisoning and procedural complications) | 1 (1)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
TENDON RUPTURE (Injury, poisoning and procedural complications) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1)
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 1 (1)
HEPATOCELLULAR CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
PANCREATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
PAPILLARY THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
TUMOUR THROMBOSIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (1)
DIZZINESS POSTURAL (Nervous system disorders) | 1 (1)
ENCEPHALOPATHY (Nervous system disorders) | 1 (1)
PARAESTHESIA (Nervous system disorders) | 1 (1)
PSYCHOMOTOR SKILLS IMPAIRED (Nervous system disorders) | 1 (1)
SYNCOPE (Nervous system disorders) | 1 (1)
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 1 (1)
AFFECT LABILITY (Psychiatric disorders) | 1 (1)
ANGER (Psychiatric disorders) | 1 (1)
INSOMNIA (Psychiatric disorders) | 1 (1)
MANIA (Psychiatric disorders) | 1 (1)
SCHIZOAFFECTIVE DISORDER (Psychiatric disorders) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1)
CALCULUS URINARY (Renal and urinary disorders) | 1 (1)
NEPHROLITHIASIS (Renal and urinary disorders) | 1 (1)
RENAL COLIC (Renal and urinary disorders) | 1 (1)
ECZEMA (Skin and subcutaneous tissue disorders) | 1 (1)
HYPERTENSION (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABT-450/r/ABT-267 Plus ABT-333 With or Without Ribavirin (RBV) (N=1596)
DIARRHOEA (Gastrointestinal disorders) | 103 (112)
NAUSEA (Gastrointestinal disorders) | 186 (200)
ASTHENIA (General disorders) | 165 (179)
FATIGUE (General disorders) | 300 (331)
HEADACHE (Nervous system disorders) | 291 (319)
INSOMNIA (Psychiatric disorders) | 179 (183)
PRURITUS (Skin and subcutaneous tissue disorders) | 199 (209)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2015-01-19): https://cdn.clinicaltrials.gov/large-docs/90/NCT02219490/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-22): https://cdn.clinicaltrials.gov/large-docs/90/NCT02219490/SAP_001.pdf